CLINICAL TRIAL: NCT03816774
Title: Effect of Adding Simethicone to a Split Regimen of Polyethylene Glycol for Bowel Preparation in a Colorectal Cancer Screening Colonoscopy Setting: an Endoscopist-blinded Randomized Controlled Trial
Brief Title: Effect of Adding Simethicone to Split-dose Polyethylene Glycol for Bowel Preparation in a Screening Colonoscopy Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Mafalda Cainé João, Principal Investigator, Portuguese Oncology Institute, Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PortugueseOIC 003
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Colo-rectal Cancer; Colonic Neoplasms
Keywords: screening colonoscopy; colo-rectal cancer; simethicone; split-dose polyethylene glycol; adequate bowel preparation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Simethicone

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG split-dose (No Intervention): Group A: PEG split dose ending 3 hours before colonoscopy
- PEG split-dose and simethicone (Active Comparator): Group B: 250mg simethicone pill 15 minutes before PEG dose on the previous evening plus 250mg simethicone pill 15 minutes before PEG dose ending 3 hours before colonoscopy
  Interventions: Drug: PEG split-dose and simethicone

INTERVENTIONS:
Drug: PEG split-dose and simethicone — Patients in active comparator arm are instructed to take 250mg simethicone pill 15 minutes before PEG dose on the previous evening plus 250mg simethicone pill 15 minutes before PEG dose ending 3 hours before colonoscopy
  Other Names: Aero-OM
  Arms: PEG split-dose and simethicone

SUMMARY:
Colonoscopy is currently accepted as the gold standard in screening, surveillance and prevention for colorectal cancer (CRC), and therefore, its quality is a major priority.

The quality of colonoscopy is greatly dependent on the quality of the bowel preparation. Standard bowel cleansing includes a low-fibre diet on the day preceding the exam and a split regimen of 4 litres of polyethylene glycol (PEG) solution.

In order to improve bowel cleansing some additional measures are available. Simethicone is an inexpensive and safe antifoaming agent that reduces the surface tension of air bubbles, theoretically presenting several benefits such as increased tolerability to the preparation, thereby improving the quality of the preparation and, secondly, adenoma detection (ADR) and cecal intubation rates (CIR). However, its role remains controversial, with some publications supporting its administration and others failing to demonstrate clear benefits.

The main aim of this study is to assess if addition of simethicone to a split-dose cleansing regimen of 4 litres of PEG improves adequate bowel preparation rate.

DETAILED DESCRIPTION:
a. Study type: Endoscopist-blinded randomized controlled trial i. Prospective inclusion of patients scheduled for a colonoscopy by nationwide CRC screening program after a positive faecal immunochemical test.

ii. Randomization by computer generated tables. iii. Allocation concealment by sealed, opaque envelopes. iv. Endoscopist-blinded: endoscopist blinded to the group allocation. v. Patient informed about its bowel cleansing regimen.

b. Selection participant method: i. Inclusion by invitation of patients aged between 50 and 74 years, inclusive, scheduled for colonoscopy by nationwide CRC screening program after a positive faecal immunochemical test. ii. Exclusion criteria for nationwide CRC screening program: previous diagnosis of CRC, presence of known genetic susceptibility syndromes related with CRC, personal history of inflammatory bowel disease, presence of gastrointestinal complaints (significant changes in gastrointestinal transit in the last 6 months or evidence of gastrointestinal bleeding), a normal colonoscopy in the last 10 years and a normal flexible sigmoidoscopy in the last 5 years. Exclusion criteria of this study also include: known or suspected gastrointestinal obstruction or perforation, toxic megacolon, major colonic resection, pregnant or at risk of becoming pregnant and lactating women, known or suspected hypersensitivity to the active or other ingredients.

c. Sample size: i. 412 (2 groups of 206 patients). ii. To improve adequate bowel preparation rate (primary outcome) from 85% (value from the investigator's own database) to 95% (target standard suggested by ESGE) and assuming a normal distribution and a power of 90% (α=0.05), the calculated sample size of each of the 2 groups was 188; allowing for a 10% dropout rate, the sample size is 206 per group (412 patients overall). Adequate bowel preparation is defined as total. Boston Bowel Preparation Scale ≥6 and ≥2 in each segment. The chosen scale is the most systematically validated and appropriate for the clinical setting.

d. Procedures and data collection methods: Form sheets filled by the endoscopist about intraprocedural measures and by the nurse about patient compliance and tolerability to the prescribed cleansing regimen.

e. Analysed variables: i. Primary outcome: adequate bowel preparation rate. ii. Secondary outcomes: ADR, CIR, compliance and tolerability related to the bowel cleansing regimen. iii. Patient characteristics and other variables: age, gender, degree of mucosal bubble reported by a comprehensive scoring used by previous studies (grade 0: no bubbles; 1: minimal or occasional bubbles (must be actively sought); 2: moderate or obviously present; 3: severe or so many bubbles that vision is obscured), withdrawal time, polyp detection rate and complications rate.

f. Statistical analysis: i. Performed using statistical software IBM SPSS Statistics, Version 25.0. Armonk, NY: IBM Corp. ii. Continuous variables are reported as mean and standard deviation or median and interquartile range, if they have normal or not normal distribution, respectively; categorical variables as absolute and relative frequency. iii. Continuous variables are compared between two groups using Student's T test if they have a normal distribution and homogeneity of variance or Mann-Whitney U if these conditions are not met. Categorical variables are compared using Pearson's X2 test or Fisher test. iv. All hypotheses are two-tailed and a P-value<0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

* consecutive patients scheduled for colonoscopy by nationwide CRC screening program after a positive faecal immunochemical test,
* signed informed consent.

Exclusion criteria:

* previous diagnosis of CRC,
* presence of known genetic susceptibility syndromes related with CRC,
* personal history of inflammatory bowel disease,
* presence of gastrointestinal complaints (significant changes in gastrointestinal transit in the last 6 months or evidence of gastrointestinal bleeding),
* a normal colonoscopy in the last 10 years and a normal flexible sigmoidoscopy in the last 5 years,
* known or suspected gastrointestinal obstruction or perforation, toxic megacolon, major colonic resection,
* pregnant or at risk of becoming pregnant and lactating women,
* known or suspected hypersensitivity to the active or other ingredients.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation rate | 1 day (during colonoscopy)
  Total BBPS ≥6 and ≥2 in each segment (ascendent, transverse, descendent), presented as percentage.

SECONDARY OUTCOMES:
Adenoma detection rate | Within 30 days from colonoscopy date
  Colonoscopies with at least one adenoma identified, presented as percentage.
Cecal intubation rate | 1 day (during colonoscopy)
  Photo documentation of the cecum is a mark for effective total colonoscopy, presented as percentage.
Compliance to the bowel cleansing regimen | 1 day (immediately before colonoscopy)
  Patient assessment, by written questionnaire, of compliance of the bowel cleansing regimen.
Tolerability to the bowel cleansing regimen:questionnaire | 1 day (immediately before colonoscopy)
  Patient assessment, by written questionnaire, of side effects of the bowel cleansing regimen.

OTHER OUTCOMES:
Degree of mucosal bubble | 1 day (during colonoscopy)
  Degree of mucosal bubble in each colonic segment (ascendent, transverse, descendent) reported by a comprehensive scoring used by previous studies (grade 0: no bubbles; 1: minimal or occasional bubbles (must be actively sought); 2: moderate or obviously present; 3: severe or so many bubbles that vision is obscured).
Withdrawal time | 1 day (during colonoscopy)
  Time spent on withdrawal of the endoscope from cecum to anal canal and inspection of the entire bowel mucosa at negative (no biopsy or therapy) colonoscopy, presented in minutes.
Polyp detection rate | Within 30 days from colonoscopy date
  Colonoscopies with a detection of at least one polyp, presented as percentage.
Patients characteristics questionnaire | 1 day (immediately before colonoscopy)
  Evaluate, using proper data collecting sheet, patient relevant data (age, gender, chronic medication, risk factors for inappropriate preparation)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Areia, PhD, Study Director — Portuguese Oncology Institute, Coimbra
Locations (1):
- Portuguese Oncology Institute - Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan C, Quintero E, Dumonceau JM, Regula J, Brandao C, Chaussade S, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Gimeno-Garcia A, Hazewinkel Y, Jover R, Kalager M, Loberg M, Pox C, Rembacken B, Lieberman D; European Society of Gastrointestinal Endoscopy. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2013 Oct;45(10):842-51. doi: 10.1055/s-0033-1344548. Epub 2013 Sep 12. PMID 24030244
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) quality improvement initiative. United European Gastroenterol J. 2017 Apr;5(3):309-334. doi: 10.1177/2050640617700014. Epub 2017 Mar 16. PMID 28507745
- [Background] Parmar R, Martel M, Rostom A, Barkun AN. Validated Scales for Colon Cleansing: A Systematic Review. Am J Gastroenterol. 2016 Feb;111(2):197-204; quiz 205. doi: 10.1038/ajg.2015.417. Epub 2016 Jan 19. PMID 26782820
- [Background] Wu L, Cao Y, Liao C, Huang J, Gao F. Systematic review and meta-analysis of randomized controlled trials of Simethicone for gastrointestinal endoscopic visibility. Scand J Gastroenterol. 2011 Feb;46(2):227-35. doi: 10.3109/00365521.2010.525714. Epub 2010 Oct 26. PMID 20977386
- [Background] Matro R, Tupchong K, Daskalakis C, Gordon V, Katz L, Kastenberg D. The effect on colon visualization during colonoscopy of the addition of simethicone to polyethylene glycol-electrolyte solution: a randomized single-blind study. Clin Transl Gastroenterol. 2012 Nov 29;3(11):e26. doi: 10.1038/ctg.2012.16. PMID 23238113
- [Background] de Leone A, Tamayo D, Fiori G, Ravizza D, Trovato C, De Roberto G, Fazzini L, Dal Fante M, Crosta C. Same-day 2-L PEG-citrate-simethicone plus bisacodyl vs split 4-L PEG: Bowel cleansing for late-morning colonoscopy. World J Gastrointest Endosc. 2013 Sep 16;5(9):433-9. doi: 10.4253/wjge.v5.i9.433. PMID 24044042
- [Background] Yoo IK, Jeen YT, Kang SH, Lee JH, Kim SH, Lee JM, Choi HS, Kim ES, Keum B, Chun HJ, Lee HS, Kim CD. Improving of bowel cleansing effect for polyethylene glycol with ascorbic acid using simethicone: A randomized controlled trial. Medicine (Baltimore). 2016 Jul;95(28):e4163. doi: 10.1097/MD.0000000000004163. PMID 27428209
- [Background] Yeh JH, Hsu MH, Tseng CM, Chen TH, Huang RY, Lee CT, Lin CW, Wang WL. The benefit of adding oral simethicone in bowel preparation regimen for the detection of colon adenoma: A systematic review and meta-analysis. J Gastroenterol Hepatol. 2019 May;34(5):830-836. doi: 10.1111/jgh.14508. Epub 2018 Nov 4. PMID 30311262
- [Background] Zhang S, Zheng D, Wang J, Wu J, Lei P, Luo Q, Wang L, Zhang B, Wang H, Cui Y, Chen M. Simethicone improves bowel cleansing with low-volume polyethylene glycol: a multicenter randomized trial. Endoscopy. 2018 Apr;50(4):412-422. doi: 10.1055/s-0043-121337. Epub 2017 Nov 13. PMID 29132175
- [Background] Pan P, Zhao SB, Li BH, Meng QQ, Yao J, Wang D, Li ZS, Bai Y. Effect of supplemental simethicone for bowel preparation on adenoma detection during colonoscopy: A meta-analysis of randomized controlled trials. J Gastroenterol Hepatol. 2019 Feb;34(2):314-320. doi: 10.1111/jgh.14401. Epub 2018 Aug 27. PMID 30069899
- [Background] Bai Y, Fang J, Zhao SB, Wang D, Li YQ, Shi RH, Sun ZQ, Sun MJ, Ji F, Si JM, Li ZS. Impact of preprocedure simethicone on adenoma detection rate during colonoscopy: a multicenter, endoscopist-blinded randomized controlled trial. Endoscopy. 2018 Feb;50(2):128-136. doi: 10.1055/s-0043-119213. Epub 2017 Oct 6. PMID 28985630
- [Background] Despacho n.o 8254/2017. Diário da República, 2.a série - N.o 183 - 21 de setembro de 2017. 2017;20788-9.
- [Background] Lazzaroni M, Petrillo M, Desideri S, Bianchi Porro G. Efficacy and tolerability of polyethylene glycol-electrolyte lavage solution with and without simethicone in the preparation of patients with inflammatory bowel disease for colonoscopy. Aliment Pharmacol Ther. 1993 Dec;7(6):655-9. doi: 10.1111/j.1365-2036.1993.tb00148.x. PMID 8161673